CLINICAL TRIAL: NCT07188090
Title: A Prospective Trial Evaluating Plerixafor-based Mobilization and Risk of Engraftment Syndrome After Autologous Hematopoietic Stem Cell Transplantation
Brief Title: Mozobil for Autologous Hematopoietic Stem Cell Transplantation
Acronym: HSCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: iRISID-2024-1641; JT 44251 (Other: JeffTrial Number)
Record Dates: First submitted 2025-09-15; First posted 2025-09-23 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Hodgkin Lymphoma; Non-hodgkin Lymphoma
Keywords: Engraftment syndrome; stem cell mobilization; autologous stem cell transplant; Plerixafor; G-CSF
MeSH Terms: conditions — Multiple Myeloma; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — plerixafor; Granulocyte Colony-Stimulating Factor; pegfilgrastim; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment with G-CSF and plerixafor for stem cell mobilization (Experimental): All patients will receive G-CSF (peg-filgrastim or filgrastim) on day -4 prior to planned peripheral blood stem cell (PBSC) collection day 0. All patients will proceed with stem cell collection on day 0. If less than 1.7 x 106 CD34+ cells/kg is collected after the first day or the target number of stem cells is not collected after two days, Plerixafor will be administered, and additional collection days will be added until the collection goal is reached.
  Interventions: Drug: Plerixafor; Drug: Gcsf

INTERVENTIONS:
Drug: Plerixafor — Plerixafor is an antagonist of chemokine receptor-4 (CXCR4) receptor that can release stem cells from the bone marrow niche into the peripheral blood circulation
  Other Names: Mozobil
Drug: Gcsf — All patients will receive G-CSF (peg-filgrastim or filgrastim) starting on day -4, prior to planned peripheral blood stem cell collection on day 0.
  Other Names: peg-filgrastim; filgrastim

SUMMARY:
This prospective trial investigates the approach of G-CSF with risk-adapted Plerixafor use for stem cell mobilization in patients undergoing autologous stem cell transplantation. Since FDA approval in 2008, Plerixafor has been combined with G-CSF to mobilize stem cells, though this regimen has been associated with a potentially higher incidence of engraftment syndrome.

The trial aims to evaluate whether using G-CSF alone, with selective use of Plerixafor, can achieve adequate stem cell collection while possibly reducing the incidence of engraftment syndrome.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label clinical trial designed to evaluate the incidence of engraftment syndrome and the efficacy of using granulocyte colonystimulating factor (G-CSF) as the primary agent for stem cell mobilization in patients undergoing autologous stem cell transplantation. The study aims to determine whether selective use of Plerixafor, administered only when necessary, can reduce the incidence of engraftment syndrome compared to a historical rate of 54%, where seventy patients with multiple myeloma or lymphoma were treated with autologous HSCT after stem cell mobilization with GCSF plus plerixafor from 2017-2021 at our institution (27).

All patients will receive G-CSF (peg-filgrastim or filgrastim) starting on day -4, prior to planned peripheral blood stem cell collection on day 0. All patients will proceed with stem cell collection on day 0. Collection will be performed via apheresis, with a collection target of approximately 3 x 106 CD34+ cells/kg of body weight. If less than 1.7 x 106 CD34+ cells/kg is collected after the first day or the target number of stem cells is not reached after two days, Plerixafor will be administered, and additional collection days will be added until the collection goal is reached. The pre-collection CD34+ cell count in peripheral blood will be measured for all participants on day 0 but will not be used to determine whether Plerixafor will be administered. The correlation between pre-collection CD34+ cell count and stem cell collection yield has been well-established (31-33).

The primary objective of the trial is to assess the incidence of engraftment syndrome, defined by clinical symptoms such as fever, rash, and capillary leakage. Incidence of engraftment syndrome will be reported separately for patients who did or did not receive Plerixafor. Secondary objectives include evaluating the efficacy of stem cell mobilization, the time to neutrophil and platelet engraftment post-transplant, the number of collection days required, length of hospital stay, patient disease response, cell composition of the collected product, and cytokine analysis.

Patients will be closely monitored throughout the mobilization and collection process, with routine blood tests performed to assess CD34+ levels, engraftment markers, and any adverse events, including engraftment syndrome. Flow cytometry will be utilized to assess the cellular composition of the collected stem cells, including measurements of CD34+ cells, mononuclear cells, lymphocyte subsets (CD3+, CD4+, CD8+), and NK cells. Additionally, cytokine levels will be measured from each subject prior to stem cell mobilization, day 10, and day 28 post-transplant. These measurements will be analyzed using appropriate assays to investigate their potential roles in the development of engraftment syndrome. The study will provide a comprehensive evaluation of whether limiting Plerixafor use can effectively reduce complications while maintaining sufficient stem cell yield for transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must meet all of the following inclusion criteria in order to be eligible to participate in the study:

  * Age ≥18 years
  * Undergoing autologous stem cell transplant for one of the following diagnoses:

    * Multiple myeloma
    * Hodgkin's lymphoma
    * Non-Hodgkin lymphoma
  * Karnofsky performance status of ≥ 60%
  * Patients must meet the TJUH BMT SOP guidelines for "Patient Criteria for Autologous HSCT" as specified below
  * Adequate organ function:

    * LVEF of ≥40%
    * Adjusted DLCO ≥45% of predicted corrected for hemoglobin
  * Adequate liver function as defined by a serum bilirubin <1.8, AST or ALT < 2.5X upper limit of normal
  * Serum creatinine ≤ 2.0 mg/dl and/or creatinine clearance of > 40 ml/min (excludes multiple myeloma patients receiving high dose Melphalan conditioning)
  * Willingness to use contraception if childbearing potential
  * Has the ability to give informed consent, or for cognitively or decisionally impaired individuals (vulnerable population), the availability of a family member or guardian to give consent and assist in the consent process
  * Life expectancy of > 12 months (exclusive of the disease for which the Auto HSCT is being performed)
  * Patients must have undergone stem cell mobilization with the combination of G- CSF or biosimilars with plerixafor or G-CSF or biosimilars alone

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Uncontrolled HIV
  * Uncontrolled bacterial infection
  * Active CNS disease
  * Pregnancy or lactation
  * Evidence of another malignancy, exclusive of a skin cancer that requires only local treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Engraftment Syndrome | 60 days post-autologous stem cell transplant
  ES will be defined as per Maiolino criteria (1) as a new fever >100.4 F without clinical or microbiological documentation of infection plus at least 1 other criteria: (1) skin rash, (2) pulmonary infiltrates in the absence of cardiac failure, pulmonary embolism, or infection, or (3) 2 or more episodes of diarrhea a day. Clinical signs of ES have to occur within 24 hours before or after the first appearance of neutrophils in the peripheral blood.

SECONDARY OUTCOMES:
Efficacy of Stem Cell Mobilization | 30 days post-autologous stem cell transplant
  To determine if G-CSF alone can successfully mobilize a sufficient number of CD34+ stem cells (approximately 3 x 106 cells/kg) in patients undergoing autologous stem cell transplantation, with Plerixafor used only when necessary. Efficacy of Stem Cell Mobilization will be analyzed using descriptive statistics and, where appropriate, survival analysis methods.
Time to Neutrophil Engraftment | Up to 90 days post-transplant
  To compare the time to engraftment of neutrophils and platelets in patients mobilized with G-CSF alone versus those requiring Plerixafor. Neutrophil engraftment is defined as ANC >500 x10e9/L x 3 days, with day of engraftment the first of the 3 days of ANC >500 x10e9/L. Platelet engraftment is defined as date platelet greater than or equal to (≥) 20 x 10e9 /L which is sustained for 3 consecutive days without a platelet transfusion within the last 7 days. Time-to-event analyses, such as Kaplan-Meier survival curves, will be used to evaluate the time to neutrophil and platelet engraftment.
Time to Platelet Engraftment | Up to 90 days post-transplant
  To compare the time to engraftment of neutrophils and platelets in patients mobilized with G-CSF alone versus those requiring Plerixafor. Neutrophil engraftment is defined as ANC >500 x10e9/L x 3 days, with day of engraftment the first of the 3 days of ANC >500 x10e9/L. Platelet engraftment is defined as date platelet greater than or equal to (≥) 20 x 10e9 /L which is sustained for 3 consecutive days without a platelet transfusion within the last 7 days. Time-to-event analyses, such as Kaplan-Meier survival curves, will be used to evaluate the time to neutrophil and platelet engraftment.
Number of Collection Days | Up to 90 days post-transplant
  To evaluate the average number of collection days needed to achieve the target CD34+ cell count, with and without Plerixafor.
Length of Hospital Stay | Up to 90 days post-transplant
  To examine whether the approach of limiting Plerixafor use influences the duration of the hospital stay for stem cell collection and transplantation.
Disease Response | Up to 90 days post-transplant
  To analyze the patient's response to treatment posttransplantation, including complete response, very good partial response, partial response, stable disease, or progressive disease.
Cell Composition | Up to 90 days post-transplant
  To investigate the composition of the collected stem cell product, particularly focusing on the percentage of CD34+ cells and other relevant immune cell populations via flow cytometry: T cell subsets (CD3+, CD4+, CD8+), B cells, natural killer (NK) cells in patients with and without Plerixafor. Cell composition data will be assessed using paired or independent t-tests, as well as ANOVA, to examine differences between groups.
Cytokine Analysis | At Baseline
  To measure and analyze cytokine levels in patients, aiming to understand the biological impact of G-CSF with or without Plerixafor on the immune response and mobilization process. Plasma levels for cytokine analysis including ESR, CRP, ferritin, interleukin (IL)-1, IL-1β, IL-2, IL-4, IL-6, interferon (IFN)-γ, tumor necrosis factor (TNF)-α, IL-12, and IL-18 will be measured from each subject prior to stem cell mobilization, day 10, and day 28 post-transplant. Cytokine analysis data will be assessed using paired or independent t-tests, as well as ANOVA, to examine differences between groups.
Cytokine Analysis | At Day 10
  To measure and analyze cytokine levels in patients, aiming to understand the biological impact of G-CSF with or without Plerixafor on the immune response and mobilization process. Plasma levels for cytokine analysis including ESR, CRP, ferritin, interleukin (IL)-1, IL-1β, IL-2, IL-4, IL-6, interferon (IFN)-γ, tumor necrosis factor (TNF)-α, IL-12, and IL-18 will be measured from each subject prior to stem cell mobilization, day 10, and day 28 post-transplant. Cytokine analysis data will be assessed using paired or independent t-tests, as well as ANOVA, to examine differences between groups.
Cytokine Analysis | At Day 28
  To measure and analyze cytokine levels in patients, aiming to understand the biological impact of G-CSF with or without Plerixafor on the immune response and mobilization process. Plasma levels for cytokine analysis including ESR, CRP, ferritin, interleukin (IL)-1, IL-1β, IL-2, IL-4, IL-6, interferon (IFN)-γ, tumor necrosis factor (TNF)-α, IL-12, and IL-18 will be measured from each subject prior to stem cell mobilization, day 10, and day 28 post-transplant. Cytokine analysis data will be assessed using paired or independent t-tests, as well as ANOVA, to examine differences between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Xia Bi, MD, MS, Principal Investigator — Xia.Bi@jefferson.edu
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States